CLINICAL TRIAL: NCT01209299
Title: Integrated Molecular Signature for the Prediction of Response to Carboplatin/Paclitaxel-Based Chemotherapy in Metastatic Melanoma
Brief Title: Biomarkers in Predicting Response to Chemotherapy in Patients With Advanced or Metastatic Melanoma Previously Treated With Carboplatin and Paclitaxel With or Without Sorafenib Tosylate
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000683300; ECOG-E2603T1
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IIIC melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — DNA Methylation; Gene Expression Profiling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: gene expression analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue in the laboratory from patients receiving carboplatin and paclitaxel with or without sorafenib tosylate may help doctors learn more about the effects of this treatment on cells. It may also help doctors understand how well patients respond to treatment.

PURPOSE: This research study is studying biomarkers in predicting response to chemotherapy in patients with advanced or metastatic melanoma previously treated with carboplatin and paclitaxel with or without sorafenib tosylate.

DETAILED DESCRIPTION:
OBJECTIVES:

* To independently correlate the gene expression and promoter methylation profiles to chemotherapy response in patients with advanced or metastatic melanoma treated with carboplatin and paclitaxel with versus without sorafenib on clinical trial ECOG-E2603.
* To develop a predictive model of chemotherapy response utilizing integrated analysis of gene expression and promoter methylation data.
* To evaluate whether the NER pathway haplotypes are associated with platinum drug resistance and survival.

OUTLINE: This is a multicenter study.

Archived paraffin-embedded tissue samples are analyzed for gene expression and promoter methylation profiles, and genes involved in the NER pathway.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of melanoma

  * Unresectable locally advanced or stage IV disease
* Received carboplatin and paclitaxel with versus without sorafenib on clinical trial ECOG-E2603
* Archived paraffin-embedded tissue samples

  * Responder (complete or partial response, or stable disease) and non-responder (disease progression or unavailable)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients enrolled on E2603 from whom samples were submitted for research
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-01-19 (Actual); Primary Completion 2012-02-19 (Actual); Study Completion 2012-02-19 (Actual)

PRIMARY OUTCOMES:
Correlation between gene expression and promoter methylation profiles to chemotherapy response | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Hussein A. Tawbi, MD, PhD, Principal Investigator — University of Pittsburgh